CLINICAL TRIAL: NCT01993693
Title: Wearable Therapeutic Ultrasound Study
Brief Title: Wearable Therapeutic Ultrasound Study for Knee Osteoarthritis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: ZetrOZ, Inc. (Industry)
Collaborators: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OA-02; 2012-1 (Other: SUNY Upstate IRB (Upstate Medical University))
Record Dates: First submitted 2013-10-24; First posted 2013-11-25 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2014-06

CONDITIONS: Knee Osteoarthritis
Keywords: knee; pain; osteoarthritis; ultrasound
MeSH Terms: conditions — Osteoarthritis, Knee; Pain; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasonic Diathermy Device (Experimental): Therapeutic ultrasound used daily.
  Interventions: Device: Ultrasonic Diathermy Device
- Sham Ultrasonic Diathermy Device (Placebo Comparator): Sham device that does not deliver ultrasound
  Interventions: Device: Sham Ultrasonic Diathermy Device

INTERVENTIONS:
Device: Ultrasonic Diathermy Device — The Ultrasonic Diathermy Device provides low intensity therapeutic ultrasound to musculoskeletal tissues and joints for the purpose of pain relief, relief of muscle spasm, treatment of joint contraction, and local increase of circulation. The device is FDA-cleared for up to 4 hours of continuous use per treatment. It is a stationary hands-free device.
  Other Names: sam
  Arms: Ultrasonic Diathermy Device
Device: Sham Ultrasonic Diathermy Device — Sham therapy delivered by Ultrasonic Diathermy Device that appears identical to active device but does not deliver ultrasound
  Other Names: Sham
  Arms: Sham Ultrasonic Diathermy Device

SUMMARY:
The purpose of this study is to evaluate the ability of a wearable therapeutic ultrasound device to reduce pain and increase mobility for subjects with knee osteoarthritis.

DETAILED DESCRIPTION:
Up to 50 million people in the U.S. suffer from some form of chronic pain, and 60% of these Americans are under 65 and have limited mobility because of knee or hip Osteoarthritis (OA). Pharmaceuticals currently dominate the treatment options due to widespread insurance coverage and convenience. However, there are a myriad of public health problems associated with analgesic use, including costs, untoward side effects, and addiction potential with opioid analgesics.

Ultrasound therapy for pain and healing has been approved by the U.S. FDA and has been in use around the globe for the last 60 years. Traditionally, ultrasound-mediated pain treatment has been delivered in clinics and has been limited to short and confined periods of 5-15 min at acoustic intensities from 1-4 W/cm2 over a course of weeks to months. Over the past decade, research has increasingly focused on lower-intensity therapeutic ultrasound (30-1000 mW/cm2) delivered over extended 1-8 hr periods. (mW = milliwatt) Recent animal studies using low-intensity therapeutic ultrasound (LITUS) have demonstrated successful inflammation reduction, reduced cartilage degeneration, and tendon and fracture healing. It is believed that using a lower-intensity ultrasonic treatment regimen over extended treatment periods works with the body's natural healing process and minimizes acoustic insult as compared with traditional, higher intensity treatments. This study proposes to evaluate clinically the first wearable low intensity ultrasound system for noninvasive treatment of arthritis pain. This technology has the potential to measurably increase the quality of life for millions of people who suffer from osteoarthritis pain by providing a safe, effective, and easy-to-use treatment.

The pilot study will test the versatile ultrasound therapy system in a clinical study that will enroll up to 60 patients with mobility-impairing knee OA. The goal of the study is to establish statistically significant data that daily 4 hour LITUS treatment decreases participant pain (Visual Analog Scale [VAS]) and improves patient mobility (measured by an accelerometer worn by each participant) over placebo devices.

ELIGIBILITY:
Individual will be included if they:

1. Have physician-diagnosed mild to moderate knee OA (OARSI atlas grades 1-2) based on fixed-flexion x-ray radiological findings for osteophytes and joint space narrowing within the past 12 months,
2. are between 35-65 years of age
3. report a frequent pain score between 4-7 (range: 0-10) during the week preceding enrollment
4. report mobility limitations because of their knee pain
5. are currently not taking any prescription pain medication other than nonsteroidal antiinflammatory drugs (NSAIDs). All pain medication taken during the study should be documented.
6. are willing not to use any cream, gel, or topical solution during the administration of treatment other than the approved ultrasound gel provided to the subject at the initiation of the study
7. are deemed appropriate by their physician to participate.

Individuals will be excluded if they:

1. cannot successfully demonstrate the ability to put on and take off the device
2. are cognitively impaired
3. have bone-on-bone crepitus
4. have severe OA or patients with little to no cartilage on the knee
5. have knee replacement or other surgical intervention
6. take variable prescription medication
7. are non-ambulatory
8. participated in a clinical trial for an investigational drug and/or agent within 30 days prior to screening
9. are currently taking neuropathic medications (ie: Neurontin, Lyrica or Topamax) and/or antidepressants (ie: Amitriptyline).

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Pain | Pain will be recorded twice a day, immediately before application of the device and then immediately after the 4 hour treatment.
  Pain will be recorded using the Visual Analogue Scale (VAS).

SECONDARY OUTCOMES:
Mobility | Mobility will be recorded logged every 5 minutes, up to 24 hours a day, by the actigraph that the subject is wearing on their wrist.
  Mobility will be measured using an actigraph that will be worn on the subject's wrist 24 hours a day.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy A. Damron, MD, Principal Investigator — SUNY Upstate Orthopedics
Locations (1):
- Upstate Orthopedics, East Syracuse, New York, United States